CLINICAL TRIAL: NCT02849808
Title: Long Term Cornea Graft Survival Study (Étude Bisontine d'Estimation de la Survie à Long Terme à Partir Des données de Suivi Internes au CHRU : Evaluation Epidémiologie Clinique)
Brief Title: Long Term Cornea Graft Survival Study
Acronym: BELIEvE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2014/230
Record Dates: First submitted 2016-07-27; First posted 2016-07-29 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Keratoconus; Fuchs' Endothelial Dystrophy
Keywords: Corneal Transplantation
MeSH Terms: conditions — Keratoconus; Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Keratoplasty patients: All patients who underwent one or more keratoplasties since january 1983.

SUMMARY:
Corneal transplantation have been performed for several decades, follow-up time in some centers now exceeds 30 years. Published long term (10 years and up) graft survivals vary considerably from center to center. These variations may be explained by differences in case-mix and surgical techniques used.

The investigators aim to better understand the factors associated with long term graft survival.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent one or more keratoplasties since january 1983.
* Age 18 and older

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent one or more keratoplasties since january 1983 at the University Hospital of Besançon
Sampling Method: Non-Probability Sample
Enrollment: 564 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2017-08-03 (Actual); Study Completion 2017-08-03 (Actual)

PRIMARY OUTCOMES:
Graft survival | 20 years

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Delbosc, MD, PhD, Principal Investigator — Opthalmology Department, CHU Besançon
Locations (1):
- Ophthalmology Departement, CHU Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bidaut-Garnier M, Monnet E, Prongue A, Montard R, Gauthier AS, Desmarets M, Mariet AS, Ratajczak C, Binda D, Saleh M, Delbosc B. Evolution of Corneal Graft Survival Over a 30-Year Period and Comparison of Surgical Techniques: A Cohort Study. Am J Ophthalmol. 2016 Mar;163:59-69. doi: 10.1016/j.ajo.2015.12.014. Epub 2015 Dec 17. PMID 26706619